CLINICAL TRIAL: NCT00578305
Title: A Randomized, Placebo Controlled, Multicenter Clinical Study Investigating Efficacy of Rituximab in the Inhibition of Joint Structural Damage Assessed by Magnetic Resonance Imaging in Patients With Rheumatoid Arthritis and Inadequate Response to Methotrexate
Brief Title: A Study of Rituximab (MabThera®/Rituxan®) in Patients With Rheumatoid Arthritis and Inadequate Response to Methotrexate
Acronym: SCORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MA21056
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methylprednisolone; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Rituximab 500 mg (Experimental): Participants received rituximab 500 mg iv on Day 1 and Day 15 of the main study. Participants received a second course of treatment on Day 1 and Day 15 after Week 24 of the main study, if they met eligibility criteria (see the Detailed Description). Participants received further treatment courses on Day 1 and Day 15 at intervals of ≥ 6 months after Week 52 in the study extension phase, if they met eligibility criteria (see the Detailed Description). Throughout the study, participants received methylprednisolone 100 mg iv prior to infusion of the investigational drug, methotrexate 7.5 to 25 mg/week orally or parenterally, and folic acid or folate ≥ 5 mg/week orally.
  Interventions: Biological: Rituximab; Drug: Methylprednisolone; Drug: Methotrexate; Drug: Folic acid or folate
- Rituximab 1000 mg (Experimental): Participants received rituximab 1000 mg iv on Day 1 and Day 15 of the main study. Participants received a second course of treatment on Day 1 and Day 15 after Week 24 of the main study, if they met eligibility criteria (see the Detailed Description). Participants received further treatment courses on Day 1 and Day 15 at intervals of ≥ 6 months after Week 52 in the study extension phase, if they met eligibility criteria (see the Detailed Description). Throughout the study, participants received methylprednisolone 100 mg iv prior to infusion of the investigational drug, methotrexate 7.5 to 25 mg/week orally or parenterally, and folic acid or folate ≥ 5 mg/week orally.
  Interventions: Biological: Rituximab; Drug: Methylprednisolone; Drug: Methotrexate; Drug: Folic acid or folate
- Placebo (Placebo Comparator): Participants received placebo intravenously (iv) on Day 1 and Day 15 of the main study. Participants received a second course of treatment on Day 1 and Day 15 after Week 24 of the main study, if they met eligibility criteria (see the Detailed Description). Participants were switched to receive rituximab 1000 mg iv on Day 1 and Day 15 at intervals of ≥ 6 months after Week 52 in the study extension phase, if they met eligibility criteria (see the Detailed Description). Throughout the study, participants received methylprednisolone 100 mg iv prior to infusion of the investigational drug, methotrexate 7.5 to 25 mg/week orally or parenterally, and folic acid or folate ≥ 5 mg/week orally.
  Interventions: Drug: Placebo; Drug: Methylprednisolone; Drug: Methotrexate; Drug: Folic acid or folate

INTERVENTIONS:
Biological: Rituximab — Rituximab was supplied as a sterile liquid for iv administration.
  Other Names: MabThera®; Rituxan®
  Arms: Rituximab 1000 mg; Rituximab 500 mg
Drug: Placebo — Placebo was supplied as a sterile liquid in single-use vials for iv administration.
  Arms: Placebo
Drug: Methylprednisolone
Drug: Methotrexate
Drug: Folic acid or folate

SUMMARY:
This 3 arm study assessed the efficacy of rituximab (MabThera®/Rituxan®) in the prevention of progression of structural joint damage in participants with active rheumatoid arthritis who had an inadequate clinical response to methotrexate. Participants were randomized to receive rituximab 500 mg intravenously (iv), rituximab 1000 mg iv, or placebo iv on days 1 and 15 every 24 weeks in the main study; all participants received concomitant methotrexate at a stable dose of 12.5-25 mg/week throughout the study. Further courses of rituximab were provided to eligible participants. Structural joint damage was assessed by magnetic resonance imaging (MRI) at baseline and at intervals during the study.

DETAILED DESCRIPTION:
There were 3 phases in the study: A 52 week long main study, a study extension phase, and a 48 week long safety follow-up phase.

The first course of treatment with placebo or rituximab was initiated on Day 1 of the 52 week long main study. A second course of treatment was initiated after Week 24, if the participant met eligibility criteria. After Week 52, eligible participants received further treatment courses at intervals ≥ 6 months in the study extension phase. No treatments were administered in the safety follow-up phase.

Participants had to meet the following eligibility criteria to receive rituximab in the study extension phase.

* Minimum of 24 weeks had passed since the first infusion of the last course of study medication.
* C-reactive protein-based Disease Activity Score 28 (DAS28-CRP) ≥ 2.6.
* Absolute neutrophil count not below 1.5 x 103/μL.
* Patient had not developed contraindications for receiving rituximab, such as:

  1. Any new or uncontrolled concomitant disease such as, but not limited to, cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine or gastrointestinal disorders.
  2. Primary or secondary immunodeficiency (history of, or currently active), including known history of HIV infection.
  3. Known active infection of any kind (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization, or treatment with iv anti-infectives within 4 weeks prior to infusion or completion of oral anti-infectives within 2 weeks prior to infusion.
* Patient was not pregnant or breast feeding.
* Patients who entered the study and were found to be hepatitis B surface antigen (HBsAg) negative, hepatitis B core antibody (HBcAb) positive, were to be negative for hepatitis B viral DNA (< 29 IU/mL) and were to have aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN) results within the last 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-80 years of age.
* Active rheumatoid arthritis for ≥ 3 months and ≤ 10 years.
* Evidence of erosive disease and/or clinical synovitis in a signal joint.
* Inadequate response to 12.5-25 mg/week methotrexate for ≥ 12 weeks.

Exclusion Criteria:

* Rheumatic autoimmune disease or inflammatory joint disease other than rheumatoid arthritis. - Any surgical procedure within 12 weeks prior to baseline.
* Previous treatment with a biologic agent or with a B cell modulating or cell depleting therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (54):
- Buenos Aires, Argentina
- Brazil (4):
  - Goiânia, Goiás
  - Curtiba, Paraná
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Canada (7):
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan
- Czechia (3):
  - Brno
  - České Budějovice
  - Prague
- Denmark (3):
  - Copenhagen
  - Hillerød
  - Hvidovre
- Tallinn, Estonia
- France (4):
  - Montpellier
  - Nice
  - Orléans
  - Toulouse
- Germany (6):
  - Bad Aibling
  - Berlin
  - Dresden
  - Erlangen
  - Halle
  - Hanover
- Greece (3):
  - Athens
  - Pátrai
  - Thessaloniki
- Riga, Latvia
- Vilnius, Lithuania
- Amsterdam, Netherlands
- Oslo, Norway
- Romania (2):
  - Bucharest
  - Cluj-Napoca
- Russia (4):
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Voronezh
- Serbia (2):
  - Belgrade
  - Niška Banja
- Spain (5):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Málaga, Malaga
  - Seville, Sevilla
  - Valencia, Valencia
- Bern, Switzerland
- Turkey (Türkiye) (4):
  - Adana
  - Ankara
  - Istanbul
  - Izmir

REFERENCES:
- [Derived] Peterfy C, Emery P, Tak PP, Ostergaard M, DiCarlo J, Otsa K, Navarro Sarabia F, Pavelka K, Bagnard MA, Gylvin LH, Bernasconi C, Gabriele A. MRI assessment of suppression of structural damage in patients with rheumatoid arthritis receiving rituximab: results from the randomised, placebo-controlled, double-blind RA-SCORE study. Ann Rheum Dis. 2016 Jan;75(1):170-7. doi: 10.1136/annrheumdis-2014-206015. Epub 2014 Oct 29. PMID 25355728

RESULTS

PARTICIPANT FLOW:
Period: Double-blind Treatment Phase
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Started | 62 | 60 | 63
Treated | 62 | 60 | 63
Completed | 59 | 56 | 49
Not Completed | 3 | 4 | 14
Period: Extension Phase
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Started | 53 | 50 | 43
Completed | 49 (Some participants completed the study in this period and did not enter the safety follow-up period.) | 49 (Some participants completed the study in this period and did not enter the safety follow-up period.) | 40 (Some participants completed the study in this period and did not enter the safety follow-up period.)
Not Completed | 4 | 1 | 3
Period: Safety Follow-up Phase
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Started | 57 (Some participants entered safety follow-up directly from the double-blind treatment period.) | 54 (Some participants entered safety follow-up directly from the double-blind treatment period.) | 54 (Some participants entered safety follow-up directly from the double-blind treatment period.)
Completed | 11 | 9 | 8
Not Completed | 46 | 45 | 46

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received any part of an infusion of the study drug during the main study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo | Total
Number analyzed (Participants) | 62 | 60 | 63 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (11.10) | 50.7 (11.65) | 50.3 (11.94) | 49.9 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 50 | 48 | 143
  Male | 17 | 10 | 15 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Magnetic Resonance Imaging (MRI) Erosion Score From Baseline to Week 24
Description: The erosion score was determined according to the Outcome Measures in Rheumatology (OMERACT) rheumatoid arthritis MRI scoring (RAMRIS) system in magnetic resonance images with and without gadolinium of 15 anatomical locations in each wrist and 10 locations in each hand in the hand and wrist with the most arthritic activity. If there was no difference in disease activity between the hands, the dominant hand was used. Images were assessed by 2 experienced blinded musculoskeletal radiologists. Each location was scored in 0.5 increments from 0 to 10 with each integer unit increment representing a 10% loss of articular bone using the following scale. 0.0=normal, no erosion; 0.5=1-5% erosion; 1.0=6-10% erosion; 1.5=11-15% erosion; 2.0=16-20% erosion; etc, up to 10.0=96-100% erosion. The individual scores were summed and normalized to a range of 0 to 100 with a higher score indicating more erosion. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All randomized participants and received any part of an infusion of study medication during the main study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 59 | 58 | 60
Units on a scale | 0.13 (2.258) | 0.39 (1.807) | 1.33 (2.235)

2. Secondary Outcome: Change in Magnetic Resonance Imaging (MRI) Erosion Score From Baseline to Weeks 12 and 52
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 60 | 62 | 63
Units on a scale
  Week 12 (n = 58, 58, 56) | 0.42 (1.693) | 0.13 (1.764) | 0.33 (4.122)
  Week 52 (n = 56, 57, 58) | 0.11 (2.623) | -0.30 (2.372) | 3.02 (4.456)

3. Secondary Outcome: Change in Magnetic Resonance Imaging (MRI) Synovitis Score From Baseline to Weeks 12, 24, and Week 52
Description: The synovitis score was determined according to the Outcome Measures in Rheumatology (OMERACT) rheumatoid arthritis MRI scoring (RAMRIS) system in magnetic resonance images of 3 wrist regions and 5 metacarpophalangeal joints in the hand and wrist with the most arthritic activity. If there was no difference in disease activity between the hands, the dominant hand was used. Images were assessed by 2 experienced blinded musculoskeletal radiologists. Each location was scored in 0.5 increments from 0 to 3 with each integer unit increment representing a 33% enhancement of the maximum volume of enhancing tissue in the synovial compartment using the following scale: 0.0=normal, no synovitis; 0.5=1-17% estimated volume of enhancement; 1.0=18-33%; 1.5=34-50%; 2.0=51-67%; 2.5=68-83%; 3.0=84-100% estimated volume of enhancement. The individual scores were summed and normalized to a range of 0 to 100 with a higher score indicating more synovitis. A negative change score indicates improvement.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Units on a scale
  Week 12 (n = 58, 58, 56) | -0.50 (1.701) | -1.15 (1.866) | -0.22 (2.050)
  Week 24 (n = 61, 59, 59) | -1.14 (1.923) | -1.81 (2.289) | 0.20 (2.257)
  Week 52 (n = 61, 59, 59) | -2.03 (2.562) | -2.73 (3.120) | -0.01 (2.700)

4. Secondary Outcome: Change in Magnetic Resonance Imaging (MRI) Osteitis Score From Baseline to Weeks 12, 24, and Week 52
Description: The osteitis score was determined according to the Outcome Measures in Rheumatology (OMERACT) rheumatoid arthritis MRI scoring (RAMRIS) system in magnetic resonance images of 15 anatomical locations in each wrist and 10 locations in each hand in the hand and wrist with the most arthritic activity. If there was no difference in disease activity between the hands, the dominant hand was used. Each location was scored in 0.5 increments from 0 to 3 with each integer unit increment representing a 33% increase in the volume of the peripheral 1 cm of original (eroded + residual) articular bone using the following scale: 0.0=normal, no osteitis; 0.5=1-17% involvement of original articular bone; 1.0=18-33%; 1.5=34-50%; 2.0=51-67%; 2.5=68-83%; 3.0=84-100% involvement of original articular bone. The individual scores were summed and normalized to a range of 0 to 100 with a higher score indicating more synovitis. A negative change score indicates improvement.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Units on a scale
  Week 12 (n = 58, 58, 56) | -2.11 (5.049) | -1.88 (5.366) | -0.14 (3.940)
  Week 24 (n = 61, 59, 59) | -2.91 (5.687) | -2.86 (5.976) | 0.07 (5.574)
  Week 52 (n = 61, 59, 59) | -4.75 (7.413) | -3.83 (6.255) | -0.22 (6.390)

5. Secondary Outcome: Percentage of Participants With no Newly Eroded Joints at Weeks 24 and 52
Description: No newly eroded joints was defined as no new erosions in joints which were scored 0 at baseline. The erosion score was determined according to the Outcome Measures in Rheumatology (OMERACT) rheumatoid arthritis MRI scoring (RAMRIS) system in magnetic resonance images with and without gadolinium of 15 anatomical locations in each wrist and 10 locations in each hand in the hand and wrist with the most arthritic activity. If there was no difference in disease activity between the hands, the dominant hand was used. Images were assessed by 2 experienced blinded musculoskeletal radiologists. Each location was scored in 0.5 increments from 0 to 10 with each integer unit increment representing a 10% loss of articular bone using the following scale. 0.0=normal, no erosion; 0.5=1-5% erosion; 1.0=6-10% erosion; 1.5=11-15% erosion; 2.0=16-20% erosion; etc, up to 10.0=96-100% erosion.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Percentage of participants
  Week 24 | 77.4 | 73.3 | 55.5
  Week 52 | 77.4 | 40 | 60.3

6. Secondary Outcome: Percentage of Participants With no Progression/no Worsening in Bone Erosion at Weeks 24 and 52
Description: There were 2 definitions of no progression/no worsening in bone erosion. A participant met the criterion for definition 1 when there was a change in the magnetic resonance imaging erosion score ≤ 0. A participant met the criteria for definition 2 when there was either (1) no change from Baseline in the MRI erosion score, (2) an increase in erosion score and the size of the increase in score was smaller than the smallest detectable change, or (3) a drop in the erosion score. The erosion score was determined according to the Outcome Measures in Rheumatology (OMERACT) rheumatoid arthritis MRI scoring (RAMRIS) system in magnetic resonance images with and without gadolinium of 15 anatomical locations in each wrist and 10 locations in each hand in the hand and wrist with the most arthritic activity. If there was no difference in disease activity between the hands, the dominant hand was used. Images were assessed by 2 experienced blinded musculoskeletal radiologists.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Percentage of participants
  Week 24 (Definition 1) | 50.0 | 51.7 | 33.3
  Week 24 (Definition 2) | 88.7 | 96.7 | 81.0
  Week 52 (Definition 1) | 48.4 | 55.0 | 27.0
  Week 52 (Definition 2) | 85.5 | 93.3 | 55.6

7. Secondary Outcome: Percentage of Participants With Improvement in Synovitis at Weeks 24 and 52
Description: There were 2 definitions of improvement in synovitis. A participant met the criterion for definition 1 when there was a drop in the magnetic resonance imaging synovitis score from Baseline > 0.5. A participant met the criterion for definition 2 when there was a drop in the magnetic resonance imaging synovitis score from Baseline > than the smallest detectable change. The synovitis score was determined according to the Outcome Measures in Rheumatology (OMERACT) rheumatoid arthritis MRI (RAMRIS) scoring system in magnetic resonance images with and without gadolinium of 15 anatomical locations in each wrist and 10 locations in each hand in the hand and wrist with the most arthritic activity. If there was no difference in disease activity between the hands, the dominant hand was used. Images were assessed by 2 experienced blinded musculoskeletal radiologists.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Percentage of participants
  Week 24 (Definition 1) | 41.9 | 56.7 | 22.2
  Week 24 (Definition 2) | 41.9 | 56.7 | 22.2
  Week 52 (Definition 1) | 54.8 | 60.0 | 25.4
  Week 52 (Definition 2) | 54.8 | 60.0 | 25.4

8. Secondary Outcome: Percentage of Participants With Improvement in Osteitis at Weeks 24 and 52
Description: There were 2 definitions of improvement in osteitis. A participant met the criterion for definition 1 when there was a drop in the magnetic resonance imaging osteitis score from Baseline > 0.5. A participant met the criterion for definition 2 when there was a drop in the magnetic resonance imaging osteitis score from Baseline > than the smallest detectable change. The osteitis score was determined according to the Outcome Measures in Rheumatology (OMERACT) rheumatoid arthritis MRI (RAMRIS) scoring system in magnetic resonance images with and without gadolinium of 15 anatomical locations in each wrist and 10 locations in each hand in the hand and wrist with the most arthritic activity. If there was no difference in disease activity between the hands, the dominant hand was used. Images were assessed by 2 experienced blinded musculoskeletal radiologists.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Percentage of participants
  Week 24 (Definition 1) | 50.0 | 51.7 | 22.2
  Week 24 (Definition 2) | 50.0 | 51.7 | 22.2
  Week 52 (Definition 1) | 58.1 | 51.7 | 27.0
  Week 52 (Definition 2) | 58.1 | 51.7 | 27.0

9. Secondary Outcome: Change From Baseline in the Disease Activity Score 28 (DAS28) at Weeks 24 and 52
Description: The DAS28 is a combined index for measuring disease activity in rheumatic arthritis (RA) and includes swollen and tender joint counts, C-reactive protein level (CRP), and general health (GH) status. The index is calculated with the following formula: DAS28 = (0.56 × √(TJC28)) + (0.28 × √(SJC28)) + (0.7 × log(CRO)) + (0.014 × GH), where TJC28 = tender joint count and SJC28 = swollen joint count, each on 28 joints, GH = a participant's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (left end = no disease activity [symptom-free and no arthritis symptoms], right end = maximum disease activity [maximum arthritis disease activity]). The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A negative change score indicates improvement.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Units on a scale
  Week 24 (n = 63, 62, 59) | -1.714 (1.2204) | -1.683 (1.0158) | -0.752 (1.1834)
  Week 52 (n = 63, 62, 59) | -2.055 (1.1844) | -1.801 (1.0443) | -0.747 (1.2557)

10. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Good, Moderate, or no Response at Weeks 24 and 52
Description: Change of the DAS28 score from Baseline was used to determine the EULAR responses. For a post-Baseline score ≤ 3.2, a change from Baseline of < -1.2 was a good response, < -0.6 to ≥ -1.2 was a moderate response, and ≥ -0.6 was no response. For a post-Baseline score > 3.2 to ≤ 5.1, a change from Baseline of < -0.6 was a moderate response and ≥ -0.6 was no response. For a post-Baseline score > 5.1, a change from Baseline < -1.2 was a moderate response and ≥ -1.2 was no response. A good response could not be achieved for post-Baseline scores > 3.2. DAS28=(0.56×√(TJC28))+(0.28×√(SJC28))+(0.7×log(CRP))+(0.014×GH), where TJC28=tender joint count (JC) and SJC28=swollen JC (28 joints), GH=a participant's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (left end=no disease activity, right end=maximum disease activity), and CRP=C-reactive protein level. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Percentage of participants
  Week 24 - No response | 33.9 | 22.0 | 58.7
  Week 24 - Moderate response | 37.1 | 42.4 | 22.2
  Week 24 - Good response | 29.0 | 35.6 | 19.0
  Week 52 (n = 63, 62, 59) - No response | 21.0 | 13.6 | 60.3
  Week 52 (n = 63, 62, 59) - Moderate response | 45.2 | 49.2 | 31.7
  Week 52 (n = 63, 62, 59) - Good response | 33.9 | 37.3 | 7.9

11. Secondary Outcome: Percentage of Participants With Low Disease Activity (Disease Activity Score 28 [DAS28] ≤ 3.2) at Weeks 24 and 52
Description: The percentage of participants who had low rheumatic arthritis disease activity at Weeks 24 and 52, as measured by a DAS28 score ≤ 3.2, is reported. DAS28 is calculated with the following formula: DAS28 = (0.56 × √(TJC28)) + (0.28 × √(SJC28)) + (0.7 × log(CRO)) + (0.014 × GH), where TJC28 = tender joint count and SJC28 = swollen joint count, each on 28 joints, GH = a participant's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (left end = no disease activity [symptom-free and no arthritis symptoms], right end = maximum disease activity [maximum arthritis disease activity]), and CRP = C-reactive protein level. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Percentage of participants
  Week 24 | 33.9 | 36.7 | 19.0
  Week 52 | 37.1 | 38.3 | 9.5

12. Secondary Outcome: Percentage of Participants in Remission Response (Disease Activity Score 28 [DAS28] < 2.6) at Weeks 24 and 52
Description: The percentage of participants in remission of their rheumatic arthritis at Weeks 24 and 52, as measured by a DAS28 score < 2.6, is reported. DAS28 is calculated with the following formula: DAS28 = (0.56 × √(TJC28)) + (0.28 × √(SJC28)) + (0.7 × log(CRO)) + (0.014 × GH), where TJC28 = tender joint count and SJC28 = swollen joint count, each on 28 joints, GH = a participant's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (left end = no disease activity [symptom-free and no arthritis symptoms], right end = maximum disease activity [maximum arthritis disease activity]), and CRP = C-reactive protein level. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Percentage of participants
  Week 24 | 21.0 | 28.3 | 12.7
  Week 52 | 25.8 | 25.0 | 7.9

13. Secondary Outcome: Percentage of Participants With an Improvement of at Least 20%, 50%, or 70% in the American College of Rheumatology (ACR) Score (ACR20/50/70) From Baseline at Weeks 24 and 52
Description: Improvement must be seen in tender and swollen joint counts (28 assessed joints; Joints were evaluated and classified as swollen or not swollen and tender or not tender based on pressure and joint manipulation upon physical examination) and in at least 3
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Percentage of participants
  Week 24 - ACR20 response | 51.6 | 51.7 | 28.6
  Week 24 - ACR50 response | 24.2 | 26.7 | 11.1
  Week 24 - ACR70 response | 11.3 | 8.3 | 1.6
  Week 52 - ACR20 response | 67.7 | 68.3 | 28.6
  Week 52 - ACR50 response | 37.1 | 35.0 | 14.3
  Week 52 - ACR70 response | 17.7 | 16.7 | 6.3

14. Secondary Outcome: Percentage of Participants Achieving a Major Clinical Response at Week 52
Description: A major clinical response was defined as an improvement of at least 70% in the American College of Rheumatology score from Baseline at Week 52. Improvement must be seen in tender and swollen joint counts (28 assessed joints) and in at least 3 of the following 5 parameters: Separate participant and physician assessments of participant disease activity in the previous 24 hours on a visual analog scale (VAS, the extreme left end of the line "no disease activity" [symptom-free and no arthritis symptoms] and the extreme right end "maximum disease activity"); participant assessment of pain in previous the 24 hours on a VAS (extreme left end of the line "no pain" and the extreme right end "unbearable pain"); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and C reactive protein level.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Percentage of participants | 6.5 | 6.7 | 1.6

15. Secondary Outcome: Correlation of Magnetic Resonance Imaging Assessments and Clinical Outcome Measures
Description: Correlation coefficients of magnetic resonance imaging erosion, synovitis, and osteitis scores and clinical outcome measures of swollen joint count (SJC), tender joint count (TJC), C-reactive protein level (CRP), erythrocyte sedimentation rate (ESR), a participant's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (GH), Disease Activity Score 28-C-reactive protein (DAS28-CRP), and Disease Activity Score 28-erythrocyte sedimentation rate (DAS28-ESR) are reported. Not all of these variables were specified as primary or secondary Outcome Measures in the study protocol and were not individually analyzed.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Number; unit: Correlation coefficient
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Correlation coefficient
  Erosion score and SJC - Week 24 | 0.341 | 0.425 | 0.446
  Erosion score and SJC - Week 52 | 0.287 | 0.234 | 0.355
  Synovitis score and SJC - Week 24 | 0.329 | 0.389 | 0.566
  Synovitis score and SJC - Week 52 | 0.168 | 0.188 | 0.574
  Osteitis score and SJC - Week 24 | 0.407 | 0.354 | 0.370
  Osteitis score and SJC - Week 52 | 0.265 | 0.192 | 0.398
  Erosion score and TJC - Week 24 | 0.364 | 0.115 | 0.298
  Erosion score and TJC - Week 52 | 0.275 | 0.067 | 0.425
  Synovitis score and TJC - Week 24 | 0.336 | 0.174 | 0.282
  Synovitis score and TJC - Week 52 | 0.142 | 0.036 | 0.421
  Osteitis score and TJC - Week 24 | 0.355 | 0.118 | 0.288
  Osteitis score and TJC - Week 52 | 0.245 | 0.048 | 0.371
  Erosion score and CRP - Week 24 | 0.185 | -0.024 | 0.006
  Erosion score and CRP - Week 52 | 0.055 | 0.098 | 0.352
  Synovitis score and CRP - Week 24 | 0.030 | 0.090 | 0.192
  Synovitis score and CRP - Week 52 | -0.077 | 0.085 | 0.311
  Osteitis score and CRP - Week 24 | -0.031 | -0.057 | 0.040
  Osteitis score and CRP - Week 52 | 0.005 | -0.010 | 0.119
  Erosion score and ESR - Week 24 | 0.321 | 0.136 | 0.197
  Erosion score and ESR - Week 52 | 0.127 | 0.188 | 0.314
  Synovitis score and ESR - Week 24 | 0.182 | 0.214 | 0.358
  Synovitis score and ESR - Week 52 | 0.185 | 0.248 | 0.360
  Osteitis score and ESR - Week 24 | 0.044 | 0.043 | 0.148
  Osteitis score and ESR - Week 52 | -0.041 | 0.116 | 0.205
  Erosion score and GH - Week 24 | 0.206 | 0.043 | 0.326
  Erosion score and GH - Week 52 | 0.063 | -0.009 | 0.316
  Synovitis score and GH - Week 24 | 0.186 | 0.221 | 0.206
  Synovitis score and GH - Week 52 | -0.026 | -0.037 | 0.286
  Osteitis score and GH - Week 24 | 0.274 | 0.122 | 0.205
  Osteitis score and GH - Week 52 | 0.106 | 0.052 | 0.136
  Erosion score and DAS28-CRP - Week 24 | 0.420 | 0.198 | 0.457
  Erosion score and DAS28-CRP - Week 52 | 0.238 | 0.127 | 0.498
  Synovitis score and DAS28-CRP - Week 24 | 0.393 | 0.349 | 0.437
  Synovitis score and DAS28-CRP - Week 52 | 0.149 | 0.150 | 0.500
  Osteitis score and DAS28-CRP - Week 24 | 0.380 | 0.209 | 0.351
  Osteitis score and DAS28-CRP - Week 52 | 0.139 | 0.143 | 0.356
  Erosion score and DAS28-ESR - Week 24 | 0.429 | 0.255 | 0.439
  Erosion score and DAS28-ESR - Week 52 | 0.244 | 0.180 | 0.473
  Synovitis score and DAS28-ESR - Week 24 | 0.398 | 0.332 | 0.438
  Synovitis score and DAS28-ESR - Week 52 | 0.198 | 0.147 | 0.514
  Osteitis score and DAS28-ESR - Week 24 | 0.353 | 0.231 | 0.353
  Osteitis score and DAS28-ESR - Week 52 | 0.108 | 0.172 | 0.356

16. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Weeks 24 and 52
Description: The HAQ-DI assesses how well the patient is able to perform 8 activities: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. The patient answers 20 questions with 1 of 4 responses with the past week as the time frame: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The highest score for any question in a category determines the category score. The total score ranges from 0 (no disability) to 3 (completely disabled). A negative change score indicates improvement.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab 500 mg | Rituximab 1000 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 63
Units on a scale
  Week 24 (n = 63, 62, 59) | -0.425 (0.5606) | -0.439 (0.4770) | -0.194 (0.5849)
  Week 52 (n = 63, 62, 59) | -0.520 (0.5873) | -0.417 (0.4450) | -0.177 (0.5943)

17. Secondary Outcome: Adverse Events (AEs), Laboratory Parameters, C-reactive Protein, ESR.
Time Frame: Throughout study
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Safety population: All participants who received any part of an infusion of the study drug during the main study.
  Some participants entered the safety follow-up period directly from the double-blind treatment period.
Groups:
- Rituximab 500 mg - Double-blind Treatment Phase; Rituximab 500 mg - Extension Phase; Rituximab 500 mg - Safety Follow-up Phase: Participants received rituximab 500 mg iv on Day 1 and Day 15 of the main study. Participants received a second course of treatment on Day 1 and Day 15 after Week 24 of the main study, if they met eligibility criteria (see the Detailed Description). Participants received further treatment courses on Day 1 and Day 15 at intervals of ≥ 6 months after Week 52 in the study extension phase, if they met eligibility criteria (see the Detailed Description). Throughout the study, participants received methylprednisolone 100 mg iv prior to infusion of the investigational drug, methotrexate 7.5 to 25 mg/week orally or parenterally, and folic acid or folate ≥ 5 mg/week orally.
- Rituximab 1000 mg - Double-blind Treatment Phase; Rituximab 1000 mg - Extension Phase; Rituximab 1000 mg - Safety Follow-up Phase: Participants received rituximab 1000 mg iv on Day 1 and Day 15 of the main study. Participants received a second course of treatment on Day 1 and Day 15 after Week 24 of the main study, if they met eligibility criteria (see the Detailed Description). Participants received further treatment courses on Day 1 and Day 15 at intervals of ≥ 6 months after Week 52 in the study extension phase, if they met eligibility criteria (see the Detailed Description). Throughout the study, participants received methylprednisolone 100 mg iv prior to infusion of the investigational drug, methotrexate 7.5 to 25 mg/week orally or parenterally, and folic acid or folate ≥ 5 mg/week orally.
- Placebo - Double-blind Treatment Phase; Placebo - Extension Phase; Placebo - Safety Follow-up Phase: Participants received placebo intravenously (iv) on Day 1 and Day 15 of the main study. Participants received a second course of treatment on Day 1 and Day 15 after Week 24 of the main study, if they met eligibility criteria (see the Detailed Description). Participants were switched to receive rituximab 1000 mg iv on Day 1 and Day 15 at intervals of ≥ 6 months after Week 52 in the study extension phase, if they met eligibility criteria (see the Detailed Description). Throughout the study, participants received methylprednisolone 100 mg iv prior to infusion of the investigational drug, methotrexate 7.5 to 25 mg/week orally or parenterally, and folic acid or folate ≥ 5 mg/week orally.
Arm/Group | Rituximab 500 mg - Double-blind Treatment Phase | Rituximab 1000 mg - Double-blind Treatment Phase | Placebo - Double-blind Treatment Phase | Rituximab 500 mg - Extension Phase | Rituximab 1000 mg - Extension Phase | Placebo - Extension Phase | Rituximab 500 mg - Safety Follow-up Phase | Rituximab 1000 mg - Safety Follow-up Phase | Placebo - Safety Follow-up Phase
Serious Adverse Events (participants affected / at risk) | 3/62 | 4/60 | 5/63 | 3/50 | 5/47 | 2/41 | 0/57 | 1/54 | 0/54
Other Adverse Events (participants affected / at risk) | 24/62 | 24/60 | 20/63 | 0/50 | 0/47 | 0/41 | 0/57 | 0/54 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 500 mg - Double-blind Treatment Phase (N=62) | Rituximab 1000 mg - Double-blind Treatment Phase (N=60) | Placebo - Double-blind Treatment Phase (N=63) | Rituximab 500 mg - Extension Phase (N=50) | Rituximab 1000 mg - Extension Phase (N=47) | Placebo - Extension Phase (N=41) | Rituximab 500 mg - Safety Follow-up Phase (N=57) | Rituximab 1000 mg - Safety Follow-up Phase (N=54) | Placebo - Safety Follow-up Phase (N=54)
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Omphalitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Omphalorrhexis (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cervix carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 500 mg - Double-blind Treatment Phase (N=62) | Rituximab 1000 mg - Double-blind Treatment Phase (N=60) | Placebo - Double-blind Treatment Phase (N=63) | Rituximab 500 mg - Extension Phase (N=50) | Rituximab 1000 mg - Extension Phase (N=47) | Placebo - Extension Phase (N=41) | Rituximab 500 mg - Safety Follow-up Phase (N=57) | Rituximab 1000 mg - Safety Follow-up Phase (N=54) | Placebo - Safety Follow-up Phase (N=54)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Immune system disorders) | 2 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 4 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.